CLINICAL TRIAL: NCT06251180
Title: A Phase Ib Study to Assess Safety and Preliminary Efficacy of Rocbrutinib in Combination with R-CHOP in Patients with Newly Diagnosed B-NHL
Brief Title: Phase Ib Study of Rocbrutinib in Combination with R-CHOP in Patients with Newly Diagnosed B-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP-168-CN301
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Escalation (Experimental): Patients with DLBCL or MCL or MZL receive Rocbrutinib（at escalating dose）+R-CHOP
  Interventions: Drug: Rocbrutinib; Biological: Rituximab; Drug: Cyclophosphamide; Drug: doxorubicin; Drug: Vincristin; Drug: Prednisone
- Dose Expansion [non-GCB DLBCL] (Experimental): Patients with non-GCB DLBCL receive Rocbrutinib（at recommended dose )+R-CHOP
  Interventions: Drug: Rocbrutinib; Biological: Rituximab; Drug: Cyclophosphamide; Drug: doxorubicin; Drug: Vincristin; Drug: Prednisone
- Dose Expansion [MCL] (Experimental): Patients with MCL receive Rocbrutinib（at recommended dose )+R-CHOP
  Interventions: Drug: Rocbrutinib; Biological: Rituximab; Drug: Cyclophosphamide; Drug: doxorubicin; Drug: Vincristin; Drug: Prednisone
- Dose Expansion [MZL] (Experimental): Patients with MZL receive Rocbrutinib（at recommended dose )+R-CHOP
  Interventions: Drug: Rocbrutinib; Biological: Rituximab; Drug: Cyclophosphamide; Drug: doxorubicin; Drug: Vincristin; Drug: Prednisone

INTERVENTIONS:
Drug: Rocbrutinib — orally once daily in a 21-day cycle for eight cycles, and as maintenance for 2 years.
  Other Names: LP-168
Biological: Rituximab — 375 mg/m2 administered intravenously once on Day 1 in a 21-day cycle for eight cycles.
  Other Names: MabThera; Rituximab Biosimilar HLX01; Rituximab biosimilar TQB2303; Henlius; Halpryza
Drug: Cyclophosphamide — 750 mg/m2 administered intravenously once on Day 1 or 2 in a 21-day cycle for six cycles.
  Other Names: CTX
Drug: doxorubicin — 50 mg/m2 administered intravenously once on Day 1 or 2 in a 21-day cycle for six cycles.
  Other Names: ADM; Adriamycin; DOX; Doxorubin hydrochloride
Drug: Vincristin — 1.4 mg/m2 administered intravenously once on Day 1 or 2 in a 21-day cycle for six cycles.
  Other Names: VCR; Vincrystine
Drug: Prednisone — 100 mg orally once on Day 1 to Day 5 in a 21-day cycle for six cycles.
  Other Names: delta.1-Cortisone; 1, 2-Dehydrocortisone

SUMMARY:
This is an open-label, multicentre Phase Ib study to evaluate the safety and preliminary efficacy of new generation Bruton Tyrosine Kinase inhibitor Rocbrutinib in combination to R-CHOP (Rituximab, Cyclophosphamide, Doxorubicin, Vincristin, Prednison) in adult patients with newly diagnosed, previously untreated B-cell Non-Hodgkin Lymphoma [Diffuse Large B-cell Lymphoma (DLBCL), Marginal Zone Lymphoma (MZL) or Mantle Cell Lymphoma (MCL)].

DETAILED DESCRIPTION:
OUTLINE:

Dose escalation portion(Part A): In the dose escalation portion of the study, the escalating doses of Rocbrutinib combined with R-CHOP may be explored, using the 3+3 principle for dose determination. If dose escalation is acceptable, and subsequently will determine the recommended Phase 2 dose.

Dose expansion portion(Part B): This will be conducted as a multicenter, open-label study, including three cohorts(Cohort 1: non-GCB DLBCL; Cohort 2: MZL; Cohort 3: MCL). Eligible subjects will receive Rocbrutinib combined with R-CHOP for 6 cycles, then Rocbrutinib plus Rituximab for 2 cycles, and followed by Rocbrutinib maintenance for 2 years.

After completion of study treatment, patients are followed up every 12 weeks for 1 year, then every 24 weeks for 4 year.

PRIMARY OBJECTIVES:

I. To evaluate the safety of Rocbrutinib in combination to R-CHOP in B-cell Non-Hodgkin Lymphoma, including the maximum tolerated dose (MTD), dose limiting toxicities(DLT), adverse events (AEs), clinically significant laboratory abnormalities.

2. To determine the recommended dose. 3. To determine the pharmacokinetic characteristics of Rocbrutinib in combination to R-CHOP.

SECONDARY OBJECTIVES:

I. To determine the overall response rate, the complete response rate, duration of remission, survival outcomes (progression free survival, event free survival, overall survival) in DLBCL/ Non-germinal Center(non-GCB) DLBCL.

2. To determine the overall response rate, the complete response rate, duration of remission, survival outcomes (progression free survival, event free survival, overall survival) in MZL.

3. To determine the overall response rate, the complete response rate, duration of remission, survival outcomes (progression free survival, event free survival, overall survival) in MCL.

ELIGIBILITY:
Inclusion Criteria:

* Participants was histopathologically diagnosed with any of the following diseases: DLBCL, MZL or MCL (if enrolled in the dose expansion phase, histological confirmation of non-GCB subtype), and have not previously received anti-tumor systemic therapy or local radiation therapy for the above diseases.
* Participants must have at least one measurable lesion.
* ECOG physical status score 0-2.
* Life expectancy ≥6 months.
* International Prognostic Index (IPI) score ≥ 2 (only participants with DLBCL in dose expansion portion).
* Adequate coagulation, liver, kidney, and hematopoietic functions：PT and APTT <1.5x ULN; serum bilirubin <1.5x ULN except in participants with Gilbert's syndrome who must have a serum bilirubin of <3x ULN, AST and ALT ≤ 3x ULN or < 5x ULN if hepatic involvement are present; serum creatinine (Scr) ≤1.5 x ULN, or calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula.; ANC≥1500/mm3, hemoglobin≥8.0 g/dL, and platelets >100,000/mm3 unless deemed related to lymphoma involvement in the bone marrow and felt potentially reversible by the treating physician.
* Women of childbearing potential must have a negative serum or urine (beta-human chorionic gonadotropin [beta-hCG]) at screening.
* Women of childbearing potential and men who are sexually active with a woman of childbearing potential must be practicing a highly effective contraceptive measures of during and after the study (90 days after the last dose of ROCBRUTINIB and 12 months after the last dose of Rituximab). Men must agree to not donate sperm during and for up to 90 days after he last dose of ROCBRUTINIB.
* Participants voluntarily enrolled and signed the informed consent form, and followed the trial treatment and visits.

Exclusion Criteria:

* Participants are allergic to Rocbrutinib or any of its excipients; Participants who are assessed by the investigator as being unable to tolerate the R-CHOP regimen.
* Participants with known central nervous system involvement with lymphoma. or diagnosis of primary central nervous system lymphoma (PCNSL) or primary mediastinal large B-cell lymphoma (PMBL).
* Participants with DLBCL had a history of indolent lymphoma such as FL or CLL (Richter's transformation), or was histopathologically comfirmed with FL (regardless of grade) coexistentially.
* Prior treatment with solid organ transplantation or hematopoietic stem cell transplantation(HSCT) ; expected HSCT during the study.
* Major surgery within 4 weeks of study entry or expected major surgery during the study.
* Prior another non-antitumor or medical instruments clinical trials within 4 weeks.
* Known bleeding diseases (such as von Willebrand's disease or hemophilia A, hemophilia B, etc.), or have bleeding tendency.
* Prior treatment with warfarin or equivalent vitamin K antagonists within 14 days; requires anticoagulation with warfarin or equivalent vitamin K antagonists.
* Prior treatment with strong/moderate CYP3A4 inhibitors within 5 days or prior foods with inhibitory effects on CYP3A4 within 3 days at screening; requires chronic treatment with moderate/strong CYP3A inhibitors or inducers, or OATP1B1/OATP1B3 sensitive substrates during the study.
* Participants with other malignancies other than the target indications of this study within the past three years.
* Prior treatment with the cumulative dose of doxorubicin ≥150 mg/m2 (or other anthracyclines at doses converted based on cumulative cardiac toxicity)
* Any serious medical condition including but not limited to uncontrolled hypertension, uncontrolled congestive heart failure or ≥Class 2 cardiac disease as defined by the New York Heart Association Functional Classification or LVEF less than 40%, uncontrolled or symptomatic arrhythmias with corrected QT interval (QTc) > 480 msec, uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, COPD, renal failure, severe hepatic disease, uncontrolled active infection, active hemorrhage.
* Known HIV infection, or syphilis infection, or hepatitis B DNA or hepatitis C RNA positive.
* Known diseases that affect drug swallowing or absorption.
* Unfit to participate in this study in the investigator's opinion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD | Up to 21 days after the initial dose
  Standard phase I 3+3 design.
Recommended Dose | Up to 1.5 years
  Recommended Dose will be determined using available safety and pharmacokinetics data upon completion of the dose escalation phase.
Incidence of AEs | From first dose of study drug to 28 days after the last dose of study drugs
  Type, frequency and severity of AEs, relationship of AEs to study treatment Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 Type, frequency and severity of AEs, relationship of AEs to study treatment Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0
Incidence of clinically significant laboratory abnormalities | From first dose of study drug to 28 days after last dose of study drug
  Clinically significant abnormalities in hematology, chemistry, coagulation and urinalysis.
Cmax of Rocbrutinib | Up to 24 hours post dose
  Maximum plasma concentration (Cmax) of Rocbrutinib.
Tmax of Rocbrutinib | Up to 24 hours post dose
  Time to maximum plasma concentration (Tmax) of Rocbrutinib.
T1/2 of Rocbrutinib | Up to 24 hours post dose
  The terminal elimination half-life (t1/2).
AUC0-t of Rocbrutinib | Up to 24 hours post dose
  Area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration of Rocbrutinib.
CL/F of Rocbrutinib | Up to 24 hours post dose
  Apparent clearance (CL/F) of Rocbrutinib.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Evey 2 cycles for 8 cycles, and followed every 3cyles for 24 months
  Assessment using the Lugano Response Criteria for Malignant Lymphoma.
Complete remission (CR) | Evey 2 cycles for 8 cycles, and followed every 3cyles for 24 months
  Assessment using the Lugano Response Criteria for Malignant Lymphoma.
Duration of Response(DOR) | Measured from the date of the first remission to the date of earliest disease progression or death, and assessed up to 5 years.
  DOR is defined as the number of days from the date of the first remission to the date of earliest disease progression or death.
Progression-Free Survival(PFS) | Measured from the date of first dose of study drug to the date of earliest disease progression or death or last visit, and assessed up to 5 years.
  PFS is defined as the number of days from the date of the first dose of study drug to the date of earliest disease progression or death.
Event-free Survival (EFS) | Measured from the date of first dose to the date of earliest evidence of disease progression, initiation of new non-protocol-specified antitumor therapy without documented progression, death, and for up to 5 years after the last subject is enrolled.
  EFS is defined as the number of days from the date of first dose to the date of earliest evidence of disease progression/relapse, or initiation of new non-protocol-specified antitumor therapy without documented progression, or death.
Overall survival (OS) | Measured from the date of date of first dose to the date of death or last visit, and for up to 5 years after the last subject is enrolled.
  OS is defined as the number of days from the date of first dose to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Cai, Ph D, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younes A, Sehn LH, Johnson P, Zinzani PL, Hong X, Zhu J, Patti C, Belada D, Samoilova O, Suh C, Leppa S, Rai S, Turgut M, Jurczak W, Cheung MC, Gurion R, Yeh SP, Lopez-Hernandez A, Duhrsen U, Thieblemont C, Chiattone CS, Balasubramanian S, Carey J, Liu G, Shreeve SM, Sun S, Zhuang SH, Vermeulen J, Staudt LM, Wilson W; PHOENIX investigators. Randomized Phase III Trial of Ibrutinib and Rituximab Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Non-Germinal Center B-Cell Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2019 May 20;37(15):1285-1295. doi: 10.1200/JCO.18.02403. Epub 2019 Mar 22. PMID 30901302
- [Background] Younes A, Thieblemont C, Morschhauser F, Flinn I, Friedberg JW, Amorim S, Hivert B, Westin J, Vermeulen J, Bandyopadhyay N, de Vries R, Balasubramanian S, Hellemans P, Smit JW, Fourneau N, Oki Y. Combination of ibrutinib with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) for treatment-naive patients with CD20-positive B-cell non-Hodgkin lymphoma: a non-randomised, phase 1b study. Lancet Oncol. 2014 Aug;15(9):1019-26. doi: 10.1016/S1470-2045(14)70311-0. Epub 2014 Jul 17. PMID 25042202